CLINICAL TRIAL: NCT02497950
Title: Evaluating the HeartMate 3™ in a Post-Market Approval Setting: The HeartMate 3 Registry (ELEVATE™)
Brief Title: HeartMate 3 ELEVATE™ Registry
Acronym: ELEVATE™
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Europe Ltd (Industry); Thoratec Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: HeartMate 3™ Registry
Record Dates: First submitted 2015-07-03; First posted 2015-07-15 (Estimated); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Cardiovascular Disease; Ventricular Dysfunction
Keywords: HeartMate 3; LVAS; LVAD; Heart-assist devices; Thoratec Corporation
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Ventricular Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HeartMate 3: This registry will include all patients that receive the HM3 LVAS in the post-market setting
  Interventions: Device: HeartMate 3

INTERVENTIONS:
Device: HeartMate 3 — Any patient that is determined to meet the HM3 commercially approved labelling indication and that is implanted with the HM3
  Other Names: HM3

SUMMARY:
Evaluate real-world experience of HeartMate 3 (HM3) in post-approval setting.

DETAILED DESCRIPTION:
The purpose of this post-market registry is to collect data and evaluate the real-world experience of the HeartMate 3 Left Ventricular Assist System (HM3 LVAS) in a post-approval setting.

ELIGIBILITY:
Inclusion:

1. Patient consented to registry data collection
2. Patient has met the HeartMate 3 commercially approved labeling indication and is implanted with the HM3.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that receive the HeartMate 3 LVAS in the post-approval setting
Sampling Method: Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD, PhD, Principal Investigator — Rigshospitalet, Denmark; Jens Garbade, MD, PhD, Principal Investigator — Gesundheit Nord Klinikverbund Bremen
Locations (26):
- AJH - Wien, Vienna, Austria
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- Germany (12):
  - Universitatsklinikum Aachen, Aachen
  - Herz- und Gefäßklinik Bad Neustadt a d Saale, Bad Neustadt an der Saale
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Medizinische Einrichtungen der Universitat Dusseldorf, Düsseldorf
  - Universitäts-Herzzentrum Freiburg, Freiberg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Herzentrum Leipzig GmbH, Leipzig
  - Universitätsklinikum Schleswig Holstein, Lübeck
  - Otto-von-Guericke-Universitat Magdeburg, Magdeburg
  - Universitätsklinikum Tübingen, Tübingen
- Sheba Medical Center, Tel Aviv, Israel
- Italy (3):
  - Ospedale San Raffaele, Milan
  - Az. Osp. San Camillo Forlanini, Roma
  - Ospedale Civile Maggiore di Verona Borgo Trento, Verona
- National Research Center for Cardiac Surgery, Astana, Kazakhstan
- Netherlands (2):
  - Erasmus MC - Thoraxcenter, Rotterdam
  - UMC Utrecht, Utrecht
- Warsaw Institute of Cardiology, Warsaw, Poland
- National Heart Centre Singapore, Singapore, Singapore
- United Kingdom (2):
  - Queen Elizabeth Hospital, Birmingham
  - Wythenshawe Hospital, Manchester

REFERENCES:
- [Derived] Zimpfer D, Gustafsson F, Potapov E, Pya Y, Schmitto J, Berchtold-Herz M, Morshuis M, Shaw SM, Saeed D, Lavee J, Heatley G, Gazzola C, Garbade J. Two-year outcome after implantation of a full magnetically levitated left ventricular assist device: results from the ELEVATE Registry. Eur Heart J. 2020 Oct 14;41(39):3801-3809. doi: 10.1093/eurheartj/ehaa639. PMID 33107561
- [Derived] Garbade J, Gustafsson F, Shaw S, Lavee J, Saeed D, Pya Y, Krabatsch T, Schmitto JD, Morshuis M, Chuang J, Zimpfer D. Postmarket Experience With HeartMate 3 Left Ventricular Assist Device: 30-Day Outcomes From the ELEVATE Registry. Ann Thorac Surg. 2019 Jan;107(1):33-39. doi: 10.1016/j.athoracsur.2018.07.092. Epub 2018 Oct 3. PMID 30291831
- [Derived] Gustafsson F, Shaw S, Lavee J, Saeed D, Pya Y, Krabatsch T, Schmitto J, Morshuis M, Chuang J, Damme L, Zimpfer D, Garbade J. Six-month outcomes after treatment of advanced heart failure with a full magnetically levitated continuous flow left ventricular assist device: report from the ELEVATE registry. Eur Heart J. 2018 Oct 1;39(37):3454-3460. doi: 10.1093/eurheartj/ehy513. PMID 30165521

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The ELEVATE study included 540 subjects of which: 482 implanted patients who provided informed consent, and 58 implanted patients had an outcome prior to having the possibility to sign the Informed Consent. For those, no patient data was collected, only duration of support and type of outcome (limited information available)
Groups:
- Elevate Full Cohort: The ELEVATE study included 540 subjects of which: 482 implanted patients who provided informed consent, and 58 implanted patients had an outcome prior to having the possibility to sign the Informed Consent. For those, no patient data was collected, only duration of support and type of outcome (limited information available)
Period: Overall Study
Arm/Group | Elevate Full Cohort
Started | 540
Completed | 208
Not Completed | 332
Not completed — Death | 209
Not completed — Transplanted | 85
Not completed — Explanted | 8
Not completed — Device Permanently Deactivated | 4
Not completed — Implanted/Exchanged to an LVAD other than HM3 | 1
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 2
Not completed — Center Did Not Participate in Long-Term FU | 4
Not completed — Refused Consent to Long-Term FU | 13

BASELINE CHARACTERISTICS:
Population: Out of the 540 enrolled patients, baseline data were not collected for 58 subjects
Groups:
- ELEVATE Consented and Implanted Patients: Patients who received HM3 and provided informed consent
Arm/Group | ELEVATE Consented and Implanted Patients
Number analyzed (Participants) | 482
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 429
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 58
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 372
  More than one race | 0
  Unknown or Not Reported | 48
Region of Enrollment [Number; unit: participants]
  Austria | 20
  Netherlands | 28
  Singapore | 6
  Czechia | 24
  Denmark | 9
  Poland | 6
  United Kingdom | 45
  Italy | 15
  Israel | 13
  Kazakhstan | 54
  Germany | 262
NYHA Class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    Class I | 5
    Class II | 2
    Class IIIA | 46
    Class IIIB | 169
    Class IV | 234
    Not provided | 26
INTERMACS Profile [Count of Participants; unit: Participants] — INTERMACS Profiles describe the Heart Failure stage of the patients:
  1. Critical cardiogenic shock
  2. Progressive decline on inotropic support
  3. Stable but inotrope dependent
  4. Resting symptoms home on oral therapy
  5. Exertion intolerant
  6. Exertion limited
  7. Advanced NYHA Class III symptom
  Participants
    1 | 43
    2 | 103
    3 | 177
    4 | 130
    5 | 9
    6 | 6
    7 | 1
    Not provided | 13
Indication [Count of Participants; unit: Participants] — The intended use of the device is either long-term (Destination Therapy), short term until a heart donor becomes available (bridge to transplant), or other.
  Participants
    Bridge to Transplant | 320
    Destination Therapy | 126
    Other Indication | 36

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Patients will be followed in the registry to 5 years post-implant or outcome (transplanted, explanted for recovery or expired), whichever occurs first.
Time Frame: Up to 5 Years post-implant
Population: The ELEVATE Study included 540 subjects of which: 482 received HM3 and provided informed consent, while 58 implanted patients had an outcome prior to having the possibility to sign the Informed Consent. For those, no patient data was collected, only duration of support and type of outcome (limited information available)
Measure: Count of Participants; unit: Participants
Groups:
- Full Cohort: The ELEVATE Full Cohort includes 540 subjects of which:
  482 implanted patients who provided informed consent 58 implanted patients who had an outcome prior having the possibility to sign the Informed Consent. For those subject no patient data was collected, only duration of support and type of outcome
Arm/Group | Full Cohort
Number analyzed (Participants) | 540
Participants | 293

2. Secondary Outcome: EuroQoL-5D-5L (EQ-5D-5L) VAS
Description: EuroQoL-5D-5L Visual Analog Score (VAS) measures self-rated health status/quality of life, with the patient indicating his/ger current status of health on a scale from 1 (extremely poor) to 100 (exceptionally good).
Time Frame: Baseline, 1, 2, 3, 4, 5 years while the patient is being supported on the HM3 LVAS
Population: Out of 540 enrolled patients, secondary outcome data were not collected for 58 patients
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- ELEVATE Patients: Out of 540 enrolled patients, secondary outcomes were not collected for 58 subjects
Arm/Group | ELEVATE Patients
Number analyzed (Participants) | 482
score on a scale
  Baseline | 35 (20)
  1 Year: number analyzed (Participants) | 282
  1 Year | 67 (18)
  2 Years: number analyzed (Participants) | 237
  2 Years | 67 (20)
  3 Years: number analyzed (Participants) | 75
  3 Years | 66 (22)
  4 Years: number analyzed (Participants) | 117
  4 Years | 65 (22)
  5 Years: number analyzed (Participants) | 124
  5 Years | 64 (20)

3. Secondary Outcome: Six Minute Walk Test (6MWT)
Description: The Six Minute Walk Test (6MWT) measures the distance that a patient can walk in a period of 6 minutes. The distance walked is measured in meters. This test measures the patients' functional status. The more meters a patient can walk over baseline indicates improvement in functional status.
Time Frame: At 5 years after implant
Population: The test was collected only if performed as per center's Standard of Care.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- ELEVATE Patients Horts: Out of 540 enrolled patients, secondary outcomes were not collected for 58 patients
Arm/Group | ELEVATE Patients Horts
Number analyzed (Participants) | 482
meters
  Baseline | 102.9 (139.5)
  1 Year: number analyzed (Participants) | 191
  1 Year | 370.7 (116.6)
  2 Years: number analyzed (Participants) | 151
  2 Years | 343.8 (127.3)
  3 Years: number analyzed (Participants) | 51
  3 Years | 356.7 (132.2)
  4 Years: number analyzed (Participants) | 63
  4 Years | 328.9 (137.7)
  5 Years: number analyzed (Participants) | 60
  5 Years | 301.2 (131.4)

4. Secondary Outcome: New York Heart Association (NYHA) Classification
Description: NYHA relates symptoms to every day activities and patients quality of life. Class 1 = no limitations on physical activity Class 2 - slight limitation of physical activity Class 3 - marked limitation of physical activity Class 4 = unable to carry out any physical activity without discomfort
Time Frame: At 5 years after implant
Population: Patients who received HM3 as either a primary implant and patients who received the HM3 or a replacement of another durable LVAD
Measure: Number; unit: participants
Groups:
- ELEVATE Patients: Out of 540 enrolled patients, secondary outcomes were not collected for 58 patients
Arm/Group | ELEVATE Patients
Number analyzed (Participants) | 482
participants
  Class I | 29
  Class II | 71
  Class III | 54
  Class IV | 3

5. Secondary Outcome: Adverse Events
Description: Frequency and incidence of pre-defined anticipated adverse event rates for patients with available data (primary implant and pump exchanges)
Time Frame: Up to 5 years post-implant
Population: The ELEVATE study included 540 subjects of which: 482 implanted patients who provided informed consent, and 58 implanted patients had an outcome prior to having the possibility to sign the Informed Consent. For those, no patient data was collected, only duration of support and type of outcome (limited information available)
Measure: Count of Participants; unit: Participants
Arm/Group | ELEVATE Patients
Number analyzed (Participants) | 482
Participants
  Arterial Non-CNS Thromboembolism | 10
  Cardiac Arrhythmias | 79
  Hemolysis | 2
  Hepatic Dysfunction | 12
  Hypertension | 12
  Major Bleeding | 155
  Major Infection | 258
  Myocardial Infarction | 3
  Neurologic Dysfunction | 73
  Pericardial Fluid Collection | 33
  Psychiatric Episode | 13
  Renal Dysfunction | 59
  Right Heart Failure | 70
  Venous Thromboembolism | 2
  Wound Dehiscence | 15
  Other Adverse Event/Adverse Device Effect | 219

6. Secondary Outcome: Device Malfunctions
Description: Number of device malfunctions reported
Time Frame: Up to 5 years post-implant
Population: as for outcome 5
Measure: Number; unit: events
Arm/Group | ELEVATE Patients
Number analyzed (Participants) | 482
events
  Thrombus: pump cover | 1
  Thrombus: inflow cannula (ingested) | 1
  Thrombus: outflow graft | 2
  Outflow graft bend relief disconnect | 1
  Outflow graft twist | 16
  Outflow graft kink | 1
  Dreiveline communication fault | 2
  Driveline damage - external | 14
  Driveline issue | 12
  Driveline disconnect causing pump stop | 3
  Driveline bend relief damage | 1
  Modular cable outer jacket tear | 1
  Controller issue | 1

7. Secondary Outcome: Reoperations
Description: Frequency and incidence of reoperations after initial implant surgery
Time Frame: Up to 5 years post-implant
Population: as for outcome 5
Measure: Number; unit: number of reoperation events
Arm/Group | ELEVATE Patients
Number analyzed (Participants) | 482
number of reoperation events | 774

8. Secondary Outcome: Rehospitalizations
Description: Frequency and incidence of rehospitalizations after initial discharge from implant surgery
Time Frame: Up to 5 years post-implant
Population: as for outcome 5
Measure: Number; unit: number of rehospitalization events
Arm/Group | ELEVATE Patients
Number analyzed (Participants) | 482
number of rehospitalization events | 1418

ADVERSE EVENTS:
Time Frame: Up to 5 years
Groups:
- ELEVATE Patients: The ELEVATE study included 540 subjects of which: 463 pts received HM3 as primary implant and 19 pts received the HM3 as a replacement of another durable LVAD. These 2 groups ( 482 pts) consist the main study population, for which complete information has been collected. In addition, 58 patients had an outcome prior to having the possibility to sign the Informed Consent. For those, no patient data was collected, only duration of support and type of outcome (limited information available)
Arm/Group | ELEVATE Patients
All-Cause Mortality (participants affected / at risk) | 209/540
Serious Adverse Events (participants affected / at risk) | 407/482
Other Adverse Events (participants affected / at risk) | 277/482
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELEVATE Patients (N=482)
Arterial Non-CNS Thromboembolism (Cardiac disorders) | 10 (11)
Cardiac Arrhythmias (Cardiac disorders) | 79 (112)
Hemolysis (Hepatobiliary disorders) | 2 (9)
Hepatic Dysfunction (Hepatobiliary disorders) | 12 (12)
Major Bleeding (Blood and lymphatic system disorders) | 155 (281)
Major Infection (Infections and infestations) | 258 (552)
Myocardial Infarction (Cardiac disorders) | 3 (3)
Neurologic Dysfunction (Nervous system disorders) | 73 (86)
Pericardial Fluid Collection (Blood and lymphatic system disorders) | 33 (38)
Psychiatric Episode (Psychiatric disorders) | 13 (14)
Renal Dysfunction (Renal and urinary disorders) | 59 (69)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 86 (95)
Right Heart Failure (Cardiac disorders) | 70 (80)
Venous Thromboembolism (Blood and lymphatic system disorders) | 2 (2)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 15 (15)
Other events (General disorders) | 219 (473)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELEVATE Patients (N=482)
Cardiac Arrhythmias (Cardiac disorders) | 53 (69)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Hepatic Dysfunction (Hepatobiliary disorders) | 8 (9)
Hypertension (Blood and lymphatic system disorders) | 23 (24)
Major Bleeding (Blood and lymphatic system disorders) | 59 (90)
Major Infection (Infections and infestations) | 166 (262)
Neurologic Dysfunction (Nervous system disorders) | 19 (20)
Pericardial Fluid Collection (Blood and lymphatic system disorders) | 3 (3)
Psychiatric Episode (Psychiatric disorders) | 20 (20)
Renal Dysfunction (Renal and urinary disorders) | 23 (27)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 17 (20)
Right Heart Failure (Cardiac disorders) | 9 (9)
Venous Thromboembolism (Blood and lymphatic system disorders) | 1 (1)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 4 (5)
Other Non Serious Events (General disorders) | 277 (826)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT02497950/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT02497950/ICF_001.pdf